CLINICAL TRIAL: NCT00688714
Title: A Randomised, Double-Blind, Placebo-Controlled Phase I Study to Assess the Tolerability, Safety, Pharmacokinetic, and Pharmacodynamic Properties of AZD6482, Alone and co-Administered With ASA, After Single Ascending Intravenous Doses to Healthy Male Subjects
Brief Title: Study to Investigate Safety and Tolerability of a Single Dose of AZD6482
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Brian Bryzinski, MD, Medical Science Director, Emerging Thrombosis, AstraZeneca R&D Mölndal, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D1700C00001
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Antiplatelet Effect
Keywords: Antiplatelet
MeSH Terms: interventions — 2-(1-(7-methyl-2-morpholin-4-yl-4-oxo-4H-pyrido(1,2-a)pyrimidin-9-yl)ethylamino)benzoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD6482
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6482 — 0,9-364,5 mg administrated through intravenous infusion over 3 hours
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
AZD6482 is a new drug substance aiming to prevent blood clots which may arise in atherosclerotic blood vessels and cause myocardial infarction or stroke. This is the first study with AZD6482 in humans. The primary aim for this study is to evaluate the safety and tolerability of AZD6482 in healthy human volunteers. How the substance is metabolised and eliminated from the body will also be studied. This will be done by comparing the effect of single ascending doses of AZD6482 to placebo (inactive substance).

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19.0 and 30.0 kg/m2, inclusive and body weight between 50.0 and 100.0 kg, inclusive
* Provision of written informed consent

Exclusion Criteria:

* Personal or family history of bleeding disorders, or reasonable suspicion of vascular malformations, including aneurysms.
* Acute illness, surgical procedure or trauma from 2 weeks before pre-entry visit until administration of investigational product or clinically significant abnormalities in clinical chemistry, haematology, faeces, urinalysis or supine BP or pulse
* Known impaired glucose intolerance or known or suspected Gilbert´s syndrome

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
General safety and tolerability including adverse events, physical examination, vital signs, ECG parameters and laboratory variables | Prior to dose, repeatedly during 24 hrs after dose and at the follow-up visit 7-10 days after.

SECONDARY OUTCOMES:
Capillary Bleeding Time, Insulin and glucose homeostasis (HoMa-Index) | Prior to dose, repeatedly during 24 hrs after dose and at the follow-up visit 7-10 days after.
Pharmacokinetics and inhibition of platelet aggregation | Prior to dose and repeatedly during 24 hrs after dose.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Hartford, MD, Principal Investigator — AstraZeneca R&D, Clinical Pharmacology Unit, Sahlgrenska University Hospital, Göteborg, Sweden; Brian Bryzinski, MD, Study Chair — AstraZeneca Wilmington, DE United States